CLINICAL TRIAL: NCT01145495
Title: A Phase II Trial of Lenalidomide (Revlimid (TM), CC-5013) (NSC #703813) Plus Rituximab in Previously Untreated Follicular Non-Hodgkin Lymphoma (NHL)
Brief Title: Lenalidomide and Rituximab in Treating Patients With Previously Untreated Stage II, Stage III, or Stage IV Follicular Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02047; NCI-2011-02047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000675161; CALGB 50803 (Other: Alliance for Clinical Trials in Oncology); CALGB-50803 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Ann Arbor Stage II Grade 1 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 1 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 2 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 2 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 3 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 3 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Grade 3 Follicular Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 3 Follicular Lymphoma
MeSH Terms: interventions — Lenalidomide; Rituximab; CT-P10

ARMS (1):
- Treatment (lenalidomide, rituximab) (Experimental): Patients receive lenalidomide PO QD on days 1-21. Treatment with lenalidomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, 15, and 22 and in weeks 13, 21, 29, and 37 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima

SUMMARY:
This phase II trial studies how well lenalidomide and rituximab work in treating patients with previously untreated stage II, stage III, or stage IV follicular non-Hodgkin lymphoma. Biological therapies, such as lenalidomide, may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Giving lenalidomide together with rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (overall and complete) to lenalidomide + rituximab in follicular non-Hodgkin lymphoma (NHL) patients who have received no prior systemic therapy.

II. To determine the time to progression after lenalidomide + rituximab in previously untreated patients with cluster of differentiation (CD)20+ follicular NHL.

SECONDARY OBJECTIVES:

I. To determine the toxicity profile of lenalidomide + rituximab therapy in previously untreated patients with CD20+ follicular NHL.

II. To establish whether the therapeutic effects of lenalidomide + rituximab combination are sufficiently promising to warrant evaluation in a subsequent randomized trial (in comparison to rituximab alone).

III. To correlate fragment crystallizable gamma (Fcg) receptor polymorphism profiling with response to lenalidomide + rituximab in previously untreated patients with follicular NHL.

IV. To determine the impact of lenalidomide on immune parameters in patients with previously untreated follicular lymphoma.

V. To determine the impact of lenalidomide on angiogenic parameters in patients with previously untreated follicular lymphoma.

VI. To correlate lymphoma-associated macrophages (LAM) and forkhead box P3 (FOXP3), granzyme B (GzB), CD10, multiple myeloma oncogene 1 (MUM1), and B-cell lymphoma 2 (BCL2) expression with response to rituximab + lenalidomide in previously untreated patients with follicular lymphoma.

VII. Determine whether immune gene signatures previously identified as prognostic factors in follicular lymphoma (FL) can be applied to paraffin-embedded tissues in rituximab treated patients; evaluate micro ribonucleic acid (RNA) signatures associated with these gene signatures and outcome; to validate immunohistochemical markers associated with outcome in FL (CD68 LAMs, FOXP3, CD10, BCL6, FOXP1, MUM1); and investigate whether markers of angiogenesis may be of value in prognosis of FL.

OUTLINE:

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21. Treatment with lenalidomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab intravenously (IV) on days 1, 8, 15, and 22 and on weeks 13, 21, 29, and 37 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 2 years and then every 6 months for up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed follicular lymphoma, World Health Organization (WHO) classification grade 1, 2, or 3a (> 15 centroblasts per high power field with centrocytes present) that is stage III, IV, or bulky (i.e., single mass >= 7 cm in any uni-dimensional measurement) stage II

  * Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies; fine needle aspirates are not acceptable for diagnosis
  * Failure to submit pathology specimens within 60 days of patient registration will be considered a major protocol violation
* Institutional flow cytometry or immunohistochemistry must confirm CD20 antigen expression
* Low or intermediate risk by Follicular Lymphoma International Prognostic Index (FLIPI): 0-2 risk factors
* No prior systemic therapy for NHL, including chemotherapy or immunotherapy (e.g., monoclonal antibody-based therapy); patients may have received involved-field radiation therapy
* No corticosteroids within two weeks prior to study entry, except for maintenance therapy for a non-malignant disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable

  * Lesions that are considered non-measurable include the following:

    * Bone lesions (lesions if present should be noted)
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Bone marrow (involvement by NHL should be noted)
* No known central nervous system (CNS) involvement by lymphoma
* Patients with human immunodeficiency virus (HIV) infection are eligible, provided they meet the following

  * No evidence of coinfection with hepatitis B or C
  * CD4+ cell count >= 400/mm^3
  * No evidence of resistant strains of HIV
  * If not on anti-HIV therapy, HIV viral load < 10,000 copies HIV RNA/mL
  * If on anti-HIV therapy, HIV viral load < 50 copies HIV RNA/mL
  * No history of acquired immune deficiency syndrome (AIDS)-defining conditions
* No evidence of active hepatitis B or C infection (i.e., no positive serology for anti-hepatitis B core [HBc] or anti-hepatitis C virus [HCV] antibodies); hepatitis B virus (HBV) seropositive patients (hepatitis B surface antigen positive [HBsAg +]) are eligible if they are closely monitored for evidence of active HBV infection by HBV deoxyribonucleic acid (DNA) testing and receive suppressive therapy with lamivudine or other HBV suppressive therapy until 6 months after the last rituximab dose
* Patients with a history of erythema multiforme, toxic epidermal necrolysis or Stevens-Johnson syndrome are not eligible
* Patients with uncontrolled seizures are not eligible
* Patients with an autoimmune disorder requires active immunosuppression are not eligible
* Non-pregnant and non-nursing; females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to registration; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* No known human anti-chimeric antibody (HACA) positivity
* Absolute neutrophil count (ANC) >= 1,000/microliter
* Platelet count >= 75,000/microliter
* Creatinine clearance >= 30 mL/min unless attributable to NHL; to be calculated by method of Cockcroft-Gault, using actual weight; maximum creatinine clearance (CrCl) 125 mL/min
* Total bilirubin =< 2 times upper limit of normal (ULN) unless attributable to NHL or Gilbert disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2022-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (91):
- United States (91):
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - AdventHealth Orlando, Orlando, Florida
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - McLeod Regional Medical Center, Florence, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017
- [Derived] Lansigan F, Barak I, Pitcher B, Jung SH, Cheson BD, Czuczman M, Martin P, Hsi E, Schoder H, Smith S, Bartlett NL, Leonard JP, Blum KA. The prognostic significance of PFS24 in follicular lymphoma following firstline immunotherapy: A combined analysis of 3 CALGB trials. Cancer Med. 2019 Jan;8(1):165-173. doi: 10.1002/cam4.1918. Epub 2018 Dec 21. PMID 30575311
- [Derived] Martin P, Jung SH, Pitcher B, Bartlett NL, Blum KA, Shea T, Hsi ED, Ruan J, Smith SE, Leonard JP, Cheson BD. A phase II trial of lenalidomide plus rituximab in previously untreated follicular non-Hodgkin's lymphoma (NHL): CALGB 50803 (Alliance). Ann Oncol. 2017 Nov 1;28(11):2806-2812. doi: 10.1093/annonc/mdx496. PMID 28945884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2010 and November 2011, 66 participants were recruited.
Pre-assignment Details: One participant did not receive protocol treatment and were dropped from all analyses.
Groups:
- Treatment (Lenalidomide, Rituximab): Patients receive oral lenalidomide (20mg) once daily on days 1-21. Treatment with lenalidomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab (375mg/m^2) IV in weeks 1, 2, 3, 4, 12, 20, 28, and 36 in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> rituximab: Given IV>
  >>
  >
  >> lenalidomide: Given orally
Period: Overall Study
Arm/Group | Treatment (Lenalidomide, Rituximab)
Started | 65
Completed | 51
Not Completed | 14
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 6
Not completed — Disease progression after respone | 2

BASELINE CHARACTERISTICS:
Population: Includes one participant did not start protocol treatment after baseline and was dropped from all analyses.
Groups:
- Treatment (Lenalidomide, Rituximab): Patients receive oral lenalidomide (20mg) once daily on days 1-21. Treatment with lenalidomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab (375mg/m^2) IV in weeks 1, 2, 3, 4, 12, 20, 28, and 36 in the absence of disease progression or unacceptable toxicity.> > rituximab: Given IV>
  > lenalidomide: Given orally
Arm/Group | Treatment (Lenalidomide, Rituximab)
Number analyzed (Participants) | 66
Age, Continuous [Median (Full Range); unit: years] | 53 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 66
Follicular Lymphoma International Prognostic Index (FLIPI) [Number; unit: participants] — Follicular Lymphoma International Prognostic Index (FLIPI) (abstracted from Solal-Céligny et al., Blood, 2004. 104(5): p. 1258-1265)>
  > Factors (1 point for each variable present): >
  * Age > 60y>
  * Ann Arbor Stage III-IV (range I-IV, with III and IV indicating highest risk)>
  * Hemoglobin level < 12 g/dL>
  * Lactate dehydrogenase (LDH) level > upper limit of normal (ULN)>
  * >= 4 nodal sites of disease>
  Risk category (factors):>
  * Low risk (0 or 1)>
  * Intermediate risk (2)>
  * High risk (> 3)
  participants
    0-1 | 21
    2 | 43
    3 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Complete Response
Description: Response is assessed by investigator according to International Working Group (IWG) criteria. Complete response requires disappearance of all evidence of disease.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide, Rituximab)
Number analyzed (Participants) | 65
Participants | 47

2. Secondary Outcome: Toxicity of Study Treatment, Assessed by the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Data will be summarized using frequency tables.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide, Rituximab)
Number analyzed (Participants) | 65
Participants
  Grade 1-2 Fatigue | 51
  Grade 1-2 Diarrhea | 24
  Grade 1-2 Rash | 21
  Grade 1-2 Febrile neutropenia | 1
  Grade 3-4 Neutropenia | 14
  Grade 3-4 Lymphopenia | 6
  Grade 3-4 Thrombocytopenia | 1
  Grade 3-4 Infection | 7
  Grade 3-4 Rash | 5

3. Secondary Outcome: Disease Progression
Description: Kaplan-Meier method will be used. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Treatment (Lenalidomide, Rituximab): Patients receive lenalidomide PO QD on days 1-21. Treatment with lenalidomide repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive rituximab IV on days 1, 8, 15, and 22 and in weeks 13, 21, 29, and 37 in the absence of disease progression or unacceptable toxicity.>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Lenalidomide: Given PO>
  > Rituximab: Given IV
Arm/Group | Treatment (Lenalidomide, Rituximab)
Number analyzed (Participants) | 65
proportion of participants
  2 Years PFS | 0.86 [0.75 to 0.93]
  3 Years PFS | 0.81 [0.69 to 0.89]
  4 Years PFS | 0.74 [0.61 to 0.86]
  5 Years PFS | 0.72 [0.58 to 0.82]

4. Secondary Outcome: Best Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide, Rituximab)
Number analyzed (Participants) | 65
Participants
  CR | 47
  PR | 15
  SD | 1
  Not evaluated | 2

ADVERSE EVENTS:
Groups:
- Treatment (Lenalidomide, Rituximab): lenalidomide: Given orally
Arm/Group | Treatment (Lenalidomide, Rituximab)
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 65/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Rituximab) (N=65)
Anemia (Blood and lymphatic system disorders) | 26 (92)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 3 (6)
Palpitations (Cardiac disorders) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 5 (16)
Sinus tachycardia (Cardiac disorders) | 1 (5)
Ear pain (Ear and labyrinth disorders) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Blurred vision (Eye disorders) | 3 (3)
Dry eye (Eye disorders) | 1 (2)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (36)
Bloating (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 19 (68)
Diarrhea (Gastrointestinal disorders) | 29 (59)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 11 (29)
Dysphagia (Gastrointestinal disorders) | 1 (3)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (9)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 3 (8)
Ileal perforation (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 8 (19)
Nausea (Gastrointestinal disorders) | 19 (48)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (12)
Chills (General disorders) | 8 (17)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 16 (50)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 56 (297)
Fever (General disorders) | 8 (9)
Flu like symptoms (General disorders) | 3 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (4)
Non-cardiac chest pain (General disorders) | 4 (11)
Pain (General disorders) | 13 (38)
Allergic reaction (Immune system disorders) | 7 (14)
Cytokine release syndrome (Immune system disorders) | 3 (3)
Serum sickness (Immune system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2)
Gum infection (Infections and infestations) | 1 (2)
Infections and infestations - Oth spec (Infections and infestations) | 4 (4)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (2)
Rash pustular (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 6 (11)
Skin infection (Infections and infestations) | 4 (9)
Soft tissue infection (Infections and infestations) | 1 (2)
Tooth infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 14 (20)
Urinary tract infection (Infections and infestations) | 5 (6)
Vaginal infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (10)
Infusion related reaction (Injury, poisoning and procedural complications) | 25 (31)
Activated partial throm time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 30 (98)
Alkaline phosphatase increased (Investigations) | 14 (38)
Aspartate aminotransferase increased (Investigations) | 22 (55)
Blood bilirubin increased (Investigations) | 11 (22)
CD4 lymphocytes decreased (Investigations) | 1 (1)
CO diffusing capacity decreased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 2 (2)
Creatinine increased (Investigations) | 6 (13)
Hemoglobin increased (Investigations) | 2 (3)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 46 (186)
Neutrophil count decreased (Investigations) | 36 (174)
Platelet count decreased (Investigations) | 30 (133)
Weight gain (Investigations) | 2 (10)
Weight loss (Investigations) | 6 (20)
White blood cell decreased (Investigations) | 41 (229)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 29 (122)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypernatremia (Metabolism and nutrition disorders) | 3 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 16 (35)
Hypoglycemia (Metabolism and nutrition disorders) | 9 (21)
Hypokalemia (Metabolism and nutrition disorders) | 11 (21)
Hyponatremia (Metabolism and nutrition disorders) | 7 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (31)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 2 (3)
Obesity (Metabolism and nutrition disorders) | 3 (24)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (41)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (35)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (6)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (4)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 5 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (24)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (18)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 6 (6)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 15 (30)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (4)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (29)
Spasticity (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (8)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 12 (37)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 6 (21)
Insomnia (Psychiatric disorders) | 12 (32)
Libido decreased (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (30)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (14)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (16)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (21)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (23)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 (76)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 10 (21)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 12 (50)
Hypotension (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (4)
Vasculitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less